CLINICAL TRIAL: NCT05481710
Title: Investigation of the Profile of Patients With Chronic Shoulder Pain: A Cross-sectional Study
Brief Title: Nociplastic Pain in Patients With Chronic Shoulder Pain
Status: Completed | Type: Observational
Sponsor: Paraskevi Bilika (Other)
Responsible Party: Sponsor-Investigator, Paraskevi Bilika, Study Director, University of Thessaly
Organization: University of Thessaly (Other)
Other Study IDs: 5
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2023-06

CONDITIONS: Chronic Shoulder Pain
Keywords: chronic pain; shoulder pain; nociplastic pain; predictors
MeSH Terms: conditions — Chronic Pain; Shoulder Pain; Nociplastic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Nociplastic Pain Criteria — All participants will be assessed with the specific nociplastic pain criteria

SUMMARY:
The aim of this study was to investigate predictors of nociplastic shoulder pain. Factors of psychological distress, functionality, fitness, quality of life, quality of sleep, functioning of the parasympathetic system, and lifestyle will be examined. Patients with nociplastic pain will be identified using the classification system proposed by the IASP.

DETAILED DESCRIPTION:
The main part of the study will include patients with chronic shoulder pain who visit the Hand Surgery-Upper Limb and Microsurgery Department of the General Hospital KAT. The measurements will be performed in one session. Once participants have been informed of the purpose and procedure of the study and given written consent, they will complete their demographics and a series of questionnaires and questions about their pain history. They will then be examined by a doctor and finally subjected to dynamometry, a functional test and two quantitative sensory tests.

ELIGIBILITY:
Inclusion Criteria:

* patients (men and women) with chronic shoulder pain (lasting more than 3 months, 3/10 Numeric Pain Rating Scale),
* aged 18-65 years
* mentally able to follow instructions or
* healthy volunteers
* aged 18-65
* who do not experience pain and have not received analgesic medication in the last trimester.

Exclusion Criteria:

* referred shoulder pain from different primary sources of pain (eg shoulder pain in women with mastectomy or stroke),
* pain manifested by movements in the neck,
* shoulder arthroplasty or fractures or dislocation of the shoulder, -
* diagnosis of chronic pain syndrome such as fibromyalgia, chronic fatigue syndrome, chronic regional pain syndrome, cancer diagnosis, osteoporosis, rheumatic inflammatory diseases,
* use of medication for neurological/psychiatric disorders,
* the presence of gastrointestinal or renal disease
* taking medication that may affect the assessment results, such as calcium channel blockers that could alter HRV,
* pregnancy or childbirth before 1 year will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The current study will include patients with chronic shoulder pain who visit the Hand Surgery-Upper Limb and Microsurgery Department of the General Hospital KAT and healthy participants who study or work at the University of Thessaly.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold (PPT) | Only one time (baseline)
  PPT will be used to assess the pain sensitivity
Conditioned Pain Modulation (CPM) | Only one time (baseline)
  CPM will be used to examine the descending inhibition of nociceptive signals
Nociplastic Pain Criteria | Only one time (baseline)
  The grading system for recognition of nociplastic pain will be used (Kosek et al. 2021).

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | Only one time (baseline)
  Pain intensity will be assessed with Numeric Pain Rating Scale. Participants will score from 0 (no pain) to 10 (the worst pain they have ever experienced).
Pain Distribution | Only one time (baseline)
  Pain location will be recorded using the Pain Distribution App (PDA) which is a self-reported tool to assess the distribution and spread of body pain areas. The PDA has demonstrated reliability.
Heart Rate Variability (HRV) | Only one time (baseline)
  HRV testing will be used to assess the function of autonomic nervous system
Range of motion | Only one time (baseline)
  Active and passive range of motion will be measured using a goniometer. It will be assessed the flexion, abduction, and external rotation. Participants will be a standing position for flexion and abduction assessment and in prone position for external rotation.
Central Sensitization Inventory (CSI) | Only one time (baseline)
  CSI wiil be used to assess the CS symptoms
Hospital Anxiety and Depression Scale (HADS) | Only one time (baseline)
  Anxiety and depression will be measured with Hospital Anxiety and Depression Scale (HADS). HADS includes 14 items, 7 for Anxiety and 7 for Depression. The overall score range 0-42 and 0-21 for the different categories. A cut-off 8/21 has been recommended.
Brief Illness Perception Questionnaire (BIPQ) | Only one time (baseline)
  BIPQ will be used to estimate the perception of pain severity
Pain Sensitivity Questionnaire (PSQ) | Only one time (baseline)
  PSQ is a self-reported tool and it will be used to assess pain sensitivity
Pain Catastrophizing Scale (PCS) | Only one time (baseline)
  PCS is a self-reported scale which estimates the catastrophization
Pain Self-Efficacy Questionnaire (PSEQ) | Only one time (baseline)
  PSEQ will be used to estimate the self-efficacy
Shoulder Pain and Disability Index (SPADI) | Only one time (baseline)
  SPADI is a self-reported questionnaire and it will be used to assess the disability
Pittsburgh Sleep Quality Index (PSQI) | Only one time (baseline)
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in adults.
Work Ability Index (WAI) | Only one time (baseline)
  WAI will be used to assess the work ability
Tampa Scale Kinesiophobia (TSK) | Only one time (baseline)
  TSK is a self-reported scale and it will be used to assess the kinesiophobia
EuroQol-5 Dimension (EQ-5D) | Only one time (baseline)
  EQ-5D will be used to assess the quality of life
3-Minute Step Test (3MST) | Only one time (baseline)
  3MST will be used to assess the cardiovascular capacity
Hand Grip | Only one time (baseline)
  Hand Grip will be used to assess the strength of forearm muscles

CONTACTS AND LOCATIONS:
Overall Officials: Paraskevi N. Bilika, Principal Investigator — University of Thessaly; Eleni V. Kapreli, Study Director — University of Thessaly
Locations (2):
- Greece (2):
  - Clinical Exercise Physiology and Rehabilitation Laboratory, Lamia, Central Greece
  - KAT Attica General Hospital, Athens

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Miller AB. The costs and benefits of breast cancer screening. Am J Prev Med. 1993 May-Jun;9(3):175-80. PMID 8347369
- See also: Psychometric properties of quantitative sensory testing focusing on healthy and patients with shoulder pain: a systematic review protocol — https://www.ijclinicaltrials.com/index.php/ijct/article/view/545